CLINICAL TRIAL: NCT03714867
Title: Use of Single Dose Pre-Operative Pregabalin for Post-Operative Analgesia in Bilateral Head and Neck Cancer Surgery: A Randomized, Double-Blinded, Placebo-Controlled Trial
Brief Title: Pre-Operative Pregabalin for Post-Operative Pain in Head and Neck Cancer Surgery
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Inability to recruit patients
Sponsor: Augusta University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1317015
Record Dates: First submitted 2018-10-19; First posted 2018-10-22 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Head and Neck Cancer; Pain, Postoperative
Keywords: head and neck cancer; analgesia; pregabalin
MeSH Terms: conditions — Head and Neck Neoplasms; Pain, Postoperative; Agnosia | interventions — Pregabalin

STUDY DESIGN:
Intervention Model Description: Intervention is single dose. Patients will be assigned to either treatment or placebo arms. No opportunity for crossing over will be present.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Patients, care providers, and investigators will all be blinded to patient group identity.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Treatment (Experimental): Treatment arm intervention consists of patients who will be administered a single enteral dose of concealed over-encapsulated Pregabalin 150mg in the pre-operative holding area. Patients will be given a post-operative regimen of 650 mg enteral acetaminophen every 6 hours and as needed oxycodone and intravenous morphine for breakthrough pain.
  Interventions: Drug: Pregabalin 150mg
- Control (Placebo Comparator): Treatment arm consists of patients who will be administered a single enteral dose of concealed over-encapsulated placebo capsules in the pre-operative holding area. Patients will be given a post-operative regimen of 650 mg enteral acetaminophen every 6 hours and as needed oxycodone and intravenous morphine for breakthrough pain.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Pregabalin 150mg — 150 mg concealed pregabalin capsule
  Other Names: Lyrica
  Arms: Treatment
Other: Placebo — Concealed placebo capsule
  Arms: Control

SUMMARY:
The purpose of this study is to evaluate and reduce pain and improve quality of life in patients being treated for head and neck cancer with primary tumor resection and bilateral neck dissections. Patients will be randomly assigned to receive either pre-operative pregabalin (Lyrica) or a placebo. Patients and investigators will be blinded to which medication patients receive, and all patients will receive the same postoperative pain medication regimen with appropriate pain treatment as needed. Patients will be asked to fill out surveys prior to surgery, while in the hospital after surgery, and at each follow-up appointment for up to 24 months.

DETAILED DESCRIPTION:
In this study, we will utilize single-dose pre-operative administration of Lyrica (pregabalin) compared to patients who will be administered a pre-operative single-dose placebo. Pregabalin is a non-narcotic GABA analogue that has been shown to be effective for the treatment of pain associated with a variety of medical conditions. Prior studies have investigated the use of single-dose pre-operative pregabalin for analgesia in acute dental, gynecologic, endoscopic thyroidectomy, and nasal septoplasty surgical pain with encouraging results demonstrating improved overall pain scores and decreased post-operative use of narcotics. Pregabalin's use for peri-operative analgesia in head and neck cancer surgery has not been evaluated.

Patients who enroll in the study will be randomly assigned by chance to receive either a single pre-operative 150 milligram dose of pregabalin (Lyrica) or placebo in the pre-operative holding area prior to proceeding with surgery. Lyrica is a non-narcotic pain medication that has been shown to promote good control of nerve-related pain in patients. Patients who agree to enroll in the study will be asked to fill out separate questionnaires to evaluate pain and quality of life preoperatively and post-operatively.

Participants will be asked to fill out four separate questionnaires to evaluate pain and quality of life pre-operatively. Patients will be administered their respective medication, either placebo or single-dose 150 milligram concealed capsule of pregabalin, by mouth in the pre-operative holding area prior to surgery. While in the hospital after surgery, patients will be given a regimen of scheduled acetaminophen 650 milligrams every 6 hours. Planned treatment of pain will include the option of requesting oxycodone on an as-needed basis every four hours and IV morphine for breakthrough pain. Surveys will be administered and collected on a daily basis while patients are in the hospital. If patients are already utilizing other non-opioid pain medications like muscle relaxers (Flexeril, baclofen, etc.), or neuropathic pain medications (Neurontin), they will be allowed to continue these medications while inpatient provided there are no changes in dosing.

Patients will be discharged home on a seven-day course of acetaminophen with as-needed oxycodone. Outcomes surveys will then be collected at each subsequent post-operative follow up. Follow up visits will occur one week after discharge, four weeks after discharge, and then every three months until completion of the two year study period.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking patients who are greater than eighteen years of age with a known diagnosis of head and neck cancer and are planned to undergo surgery with bilateral neck dissections will be eligible for this study.

Exclusion Criteria:

* Patients with a history of preoperative narcotic use for conditions unrelated to their head and neck cancer will be excluded.
* Patients younger than eighteen years of age, patients with previous severe adverse reaction to pregabalin (Lyrica), patients with a history of angioedema, and pregnant patients will be excluded from this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-03-22 (Actual); Primary Completion 2020-07-07 (Actual); Study Completion 2020-07-07 (Actual)

PRIMARY OUTCOMES:
Brief Pain Inventory | 2 years
  Validated head and neck cancer pain scale

SECONDARY OUTCOMES:
Defense and Veterans Pain Rating Scale | 2 years
  Non-validated pain scale in head and neck cancer
University of Washington Quality of Life Scale Version 4 (UW-QOL-4) | 2 years
  Validated quality of life scale in head and neck cancer
EuroQol 5D-5L | 2 years
  Non-validated quality of life scale in head and neck cancer
Inpatient morphine equivalents | 1-7 days or longer depending on length of stay
  Cumulative inpatient narcotic consumption

CONTACTS AND LOCATIONS:
Overall Officials: James K Byrd, MD, Principal Investigator — Augusta University
Locations (1):
- Augusta University Department of Otolaryngology-Head and Neck Surgery, Augusta, Georgia, United States

REFERENCES:
- [Background] Hwang SH, Park IJ, Cho YJ, Jeong YM, Kang JM. The efficacy of gabapentin/pregabalin in improving pain after tonsillectomy: A meta-analysis. Laryngoscope. 2016 Feb;126(2):357-66. doi: 10.1002/lary.25636. Epub 2015 Sep 25. PMID 26404562
- [Background] Oltman J, Militsakh O, D'Agostino M, Kauffman B, Lindau R, Coughlin A, Lydiatt W, Lydiatt D, Smith R, Panwar A. Multimodal Analgesia in Outpatient Head and Neck Surgery: A Feasibility and Safety Study. JAMA Otolaryngol Head Neck Surg. 2017 Dec 1;143(12):1207-1212. doi: 10.1001/jamaoto.2017.1773. PMID 29049548
- [Background] Sanders JG, Cameron C, Dawes PJD. Gabapentin in the Management of Pain following Tonsillectomy: A Randomized Double-Blind Placebo-Controlled Trial. Otolaryngol Head Neck Surg. 2017 Nov;157(5):781-790. doi: 10.1177/0194599817719883. Epub 2017 Jul 25. PMID 28741425
- [Background] Ogawa S, Arakawa A, Hayakawa K, Yoshiyama T. Pregabalin for Neuropathic Pain: Why Benefits Could Be Expected for Multiple Pain Conditions. Clin Drug Investig. 2016 Nov;36(11):877-888. doi: 10.1007/s40261-016-0423-x. PMID 27448285
- [Background] Moore RA, Straube S, Wiffen PJ, Derry S, McQuay HJ. Pregabalin for acute and chronic pain in adults. Cochrane Database Syst Rev. 2009 Jul 8;(3):CD007076. doi: 10.1002/14651858.CD007076.pub2. PMID 19588419
- [Background] Ben-Menachem E. Pregabalin pharmacology and its relevance to clinical practice. Epilepsia. 2004;45 Suppl 6:13-8. doi: 10.1111/j.0013-9580.2004.455003.x. PMID 15315511
- [Background] Sabatowski R, Galvez R, Cherry DA, Jacquot F, Vincent E, Maisonobe P, Versavel M; 1008-045 Study Group. Pregabalin reduces pain and improves sleep and mood disturbances in patients with post-herpetic neuralgia: results of a randomised, placebo-controlled clinical trial. Pain. 2004 May;109(1-2):26-35. doi: 10.1016/j.pain.2004.01.001. PMID 15082123
- [Background] Liebana-Hermoso S, Manzano-Moreno FJ, Vallecillo-Capilla MF, Olmedo-Gaya MV. Oral pregabalin for acute pain relief after cervicofacial surgery: a systematic review. Clin Oral Investig. 2018 Jan;22(1):119-129. doi: 10.1007/s00784-017-2272-2. Epub 2017 Nov 3. PMID 29101547
- [Background] Kim SY, Jeong JJ, Chung WY, Kim HJ, Nam KH, Shim YH. Perioperative administration of pregabalin for pain after robot-assisted endoscopic thyroidectomy: a randomized clinical trial. Surg Endosc. 2010 Nov;24(11):2776-81. doi: 10.1007/s00464-010-1045-7. Epub 2010 Apr 8. PMID 20376496
- [Background] Ringash J, Bernstein LJ, Cella D, Logemann J, Movsas B, Murphy B, Trotti A, Wells N, Yueh B, Ridge J. Outcomes toolbox for head and neck cancer research. Head Neck. 2015 Mar;37(3):425-39. doi: 10.1002/hed.23561. Epub 2015 Jan 22. PMID 24318166